CLINICAL TRIAL: NCT05540431
Title: Evaluation of Protective Effect of Activated Charcoal and Probiotic Against Progression of Chronic Kidney Disease
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Waleed Khaild Rahman Kareem Al-kabi (Other)
Responsible Party: Sponsor-Investigator, Waleed Khaild Rahman Kareem Al-kabi, Evaluation of Protective Effect of Activated Charcoal and Probiotic Against Progression of Chronic Kidney Disease, Kufa University
Organization: Kufa University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Uremic toxin in CKD
Record Dates: First submitted 2022-09-02; First posted 2022-09-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Uremic Toxin
Keywords: Indoxyl sulfate
MeSH Terms: interventions — Charcoal; Probiotics

STUDY DESIGN:
Intervention Model Description: Interventional (clinical trial)
Masking Description: None (Open Label)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Activated charcoal (Other): 1st group
  Oral activated charcoal
  20 to 25 patient with CKD will receive standard care plus Activated charcoal capsule (charconut) three times dialy for six weeks.
  Interventions: Drug: Activated Charcoal
- Probiotic (Other): 2nd group
  Oral probiotic
  20 to 25 patient with CKD will receive standard care plus Probiotic tablet twice dialy for six weeks.
  Interventions: Dietary Supplement: Probiotic
- Control group (Other): 3rd group
  Control group
  20 to 25 patient with CKD will receive standard care only for six weeks.
  Interventions: Other: No intervention

INTERVENTIONS:
Drug: Activated Charcoal — RCT
  Arms: Activated charcoal
Dietary Supplement: Probiotic — RCT
  Arms: Probiotic
Other: No intervention — RCT
  Arms: Control group

SUMMARY:
Investigate the nephroprotective effect of Activated Charcoal and Probiotic in limiting the progression of renal impairment in patients with chronic kidney disease and improving of renal function test and phosphate level.

Condition or disease:

chronic kidney disease

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is characterized by a gradual decrease in the glomerular filtration rate (GFR) and proteinuria. CKD is a global health problem, and its incidence has been increasing. The estimated global prevalence of CKD is 8-14%. When kidney function deteriorates gradually, many metabolites accumulate in the body. These accumulated substances, termed as uremic toxins (UTs), can result in adverse pathophysiological outcomes. UTs can affect multiple organs and cause renal fibrosis, vascular calcification, anemia, peripheral arterial disease, adynamic bone disease, adipocyte dysfunction with insulin resistance, impaired immune system, and uremic pruritus.

The pathophysiological mechanisms through which UTs cause multiple organ damage are complex and not completely understood. These mechanisms may include inflammation, reactive oxidative stress, cellular transdifferentiation, impaired mitochondria function, intestinal barrier destruction, and changes in intestinal microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age more than 18 years old;
* Patients with CKD;
* Both genders will be included.

Exclusion Criteria:

* Patient with age less than 18 years old;
* Inability or rejection to take activated charcoal or probiotic;
* Clinically unstable;
* Pregnant;
* Unlikely to adhere to study procedure (eg. due to cognitive limitations, severe psychiatric disorder or alcoholism).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-25 (Estimated); Primary Completion 2023-09-20 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
Improving of blood urea | Baseline to 6 week
  The concentration of blood urea(mmol/L),dL) ) in all blood samples
Indoxyl sulfate assay | Baseline to 6 week
  The concentration of human indoxyl sulfates level by elisa technique in the subjects' blood samples
Improving of serum creatinine mg/dL | Baseline to 6 week
  The concentration of serum creatinine(mg/dL) in all blood sample

SECONDARY OUTCOMES:
Nutrition status | Baseline to 6 week
  The concentration of albumin(g/dL) in the subjects' blood samples

CONTACTS AND LOCATIONS:
Locations (1):
- Waleed Khaild Rahman Alkabi, Al-diwanyia, Iraq

REFERENCES:
- [Background] Saran R, Robinson B, Abbott KC, Agodoa LYC, Bhave N, Bragg-Gresham J, Balkrishnan R, Dietrich X, Eckard A, Eggers PW, Gaipov A, Gillen D, Gipson D, Hailpern SM, Hall YN, Han Y, He K, Herman W, Heung M, Hirth RA, Hutton D, Jacobsen SJ, Jin Y, Kalantar-Zadeh K, Kapke A, Kovesdy CP, Lavallee D, Leslie J, McCullough K, Modi Z, Molnar MZ, Montez-Rath M, Moradi H, Morgenstern H, Mukhopadhyay P, Nallamothu B, Nguyen DV, Norris KC, O'Hare AM, Obi Y, Park C, Pearson J, Pisoni R, Potukuchi PK, Rao P, Repeck K, Rhee CM, Schrager J, Schaubel DE, Selewski DT, Shaw SF, Shi JM, Shieu M, Sim JJ, Soohoo M, Steffick D, Streja E, Sumida K, Tamura MK, Tilea A, Tong L, Wang D, Wang M, Woodside KJ, Xin X, Yin M, You AS, Zhou H, Shahinian V. US Renal Data System 2017 Annual Data Report: Epidemiology of Kidney Disease in the United States. Am J Kidney Dis. 2018 Mar;71(3 Suppl 1):A7. doi: 10.1053/j.ajkd.2018.01.002. No abstract available. PMID 29477157